CLINICAL TRIAL: NCT02666144
Title: Comparison of Optic Nerve Head and Retinal Nerve Fiber Layer Parameters Derived From Two Different Methods of Scan Alignment
Status: Completed | Type: Observational
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: S-2015-6
Record Dates: First submitted 2016-01-19; First posted 2016-01-28 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Glaucoma
  Interventions: Device: Spectralis OCT
- Normal
  Interventions: Device: Spectralis OCT

INTERVENTIONS:
Device: Spectralis OCT — Measurement of structural parameters of the optic nerve head (ONH), in particular, the neuroretinal rim of the ONH, and the peripapillary retinal nerve fiber layer.

SUMMARY:
This prospective, monocentric, non-invasive clinical study is designed to measure normal structural parameters of the optic nerve head, the peripapillary retinal nerve fiber layer, and the macula using the Heidelberg Spectralis OCT device. This study is conducted in normal, healthy volunteers and glaucoma patients. The main goal of the study is to provide an analysis of the comparability of these parameters between two different software versions and their respective method of scan centration on the optic disc center. The study will include at least 40 eyes of 40 subjects; 20 normal, healthy subjects and 20 glaucoma patients. All subjects will undergo Spectralis OCT imaging, biometric and ophthalmoscopic examination, and visual field testing in one single visit. Total study duration (first patient first visit to last patient last visit) is anticipated to be approximately 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to undergo the test procedures, give consent, and to follow instructions
* Subjects that understand the nature of the trial
* Signed informed consent
* Age : 18 years or older
* For "normal subjects", "normal" means, there is no reason that would prevent imaging of the eye, therefore:
* Self-reported healthy eyes without prior intraocular surgery (except cataract surgery and laser in situ keratomileusis) and without clinically significant vitreal, retinal or choroidal diseases, diabetic retinopathy, or disease of the optic nerve (e.g. impacting central VA or RNFLT measurements as determined by the expertise of the investigator)
* Visual field GHT within normal limits
* For "glaucoma subjects": Early to advanced glaucoma according to existing medical charts and visual field GHT outside normal limits on at least two occasions during the testing.
* Refraction between +6 and -6 diopters spherical equivalent and astigmatism ≤ 2 diopters
* When both eyes are eligible, one randomly selected eye will be evaluated in the analysis

Exclusion Criteria:

* Vulnerable subjects (as defined in ISO 14155 GCP)with the exception of employees of the site, and , if applicable, students of the respective university. Staff that is directly involved in the study is excluded from participation.
* subjects unable to read or write
* Unreliable visual field. The reliability indices should be used as guide as well as the perimetrist's notes.
* Unusable disc stereo photos.
* Inability to undergo the tests.
* Insufficient quality of Spectralis OCT images (this is not determined until after Spectralis OCT examination, and is an unusual circumstance).

Minimum requirements are:

* Retina completely included in image frame,
* Quality Score ≥ 20 in the stored ART mean images, and
* For ONH-R scan: Center position error ≤ 100 μm.
* Note: Inability of a subject to perform one of the two scan patterns or insufficient image quality in one scan pattern does not exclude the subject or eye from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 eyes of 20 normal healthy subjects and 20 eyes of 20 glaucoma patients, both genders approx. equally.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Agreement (Differences) of peripapillary retinal nerve fiber layer thickness | 4 weeks
  Agreement (Differences) of peripapillary retinal nerve fiber layer thickness in sectors temporal, nasal, nasal superior, nasal inferior, temporal superior and temporal inferior when measured with two different software versions.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Dul, OD, Principal Investigator — State University of New York College of Optometry